CLINICAL TRIAL: NCT05440734
Title: Sleep and Circadian Rhythms in Men and Women - Protocol 4
Brief Title: Exogenous Melatonin in Postmenopausal Women with Insomnia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Diane B. Boivin, Director, Centre for Study and Treatment of Circadian Rhythms, Douglas Mental Health University Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-175
Record Dates: First submitted 2022-06-17; First posted 2022-07-01 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Insomnia
Keywords: menopause; aging; melatonin; circadian rhythms; sleep; alertness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Randomized crossover placebo-controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The nature of the treatment (melatonin vs placebo) will only be unrevealed when the key parameters have been determined (e.g, PSG sleep scoring, alertness levels, vasomotor symptoms, adverse effects, hormone levels).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Experimental): 2 mg oral tablet, melatonin slow release formulation, 1x 60 min before bedtime for 15 days
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): 2 mg oral tablet, 1x 60 min before bedtime for 15 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — 2 Mg Oral Tablet, slow release
  Arms: Melatonin
Drug: Placebo — placebo pill identical to the treatment pill
  Arms: Placebo

SUMMARY:
The aim of the study is to assess the effect of exogenous melatonin, 2 mg SR, 60 minutes before bedtime for 15 days, on the sleep and circadian rhythms of postmenopausal women with insomnia in a randomized crossover placebo-controlled study.

DETAILED DESCRIPTION:
Eligible participants will be contacted by the research team to provide informed consent for the study. Once the screening phase is completed, they will be ready to start the study consisting of:

A) a ~2-week ambulatory phase at home with melatonin or placebo treatment; B) a 2-week wash-out period; C) same as A with the opposite treatment;

Part A: The research project will start with a 16-day ambulatory data-collection period during which participants will receive either melatonin or a placebo. They will take 2 mg of exogenous melatonin in a slow release formulation (or placebo), 60 mins prior to bedtime for 15 days. Participants will be instructed to go to bed at a regular time and stay in darkness for 8 consecutive hours each night, trying to sleep.

Part B: Throughout this period, all participants will stop taking their melatonin/placebo pills. After at least 2 weeks, they will prepare to participate to the other study condition.

Parts C: Repetition of Ambulatory phase 1 (Part A) except that participants who received the active treatment will now receive placebo and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* Insomniac women will meet the diagnostic criteria for persistent insomnia as described in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). They will report subjective sleep onset and/or maintenance difficulties associated with impaired daytime functioning at least 3 times a week, for at least 3 months. Sleep disturbances will be coincident with the onset of the menopausal transition.
* Postmenopausal women will have amenorrhea for at least 12 months.
* Participants will be drug-free at the time of study, and will have a history of only moderate or no use of coffee (≤3 cups/day), tobacco (≤ 10 cigarettes/day), alcohol (≤ 15 drinks/week), or other compounds.

Exclusion Criteria:

* Evidence of psychopathology on the Structured Clinical Interview for DSM-5, the Seasonal Pattern Assessment Questionnaire, the Beck Depression Inventory, and the Spielberger State Trait Anxiety Inventory.
* A history of prior gynecological pathology or medical condition that can affect the study results, including bilateral oophorectomy or endocrinopathy, and will not have used investigational drugs within 4 weeks of the study.
* A history of night work or transmeridian travel (across >2 time zones) in the 2 months prior to the study.
* Evidence of sleep apnea (apnea/hypopnea index > 15 per hour of sleep) or restless legs, or periodic limb movements during sleep (number of PLMs >15 per hour of sleep).

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in sleep duration | Change from baseline sleep duration at treatment day 15
  Sleep recorded with a portable device
Change in wake after sleep onset | Change from baseline sleep duration at treatment day 15
  Sleep recorded with a portable device
Change in sleep efficiency | Change from baseline sleep duration at treatment day 15
  Sleep recorded with a portable device
Urinary 6-sulfatoxy-melatonin levels | During sleep periods during the last 3 days of each treatment phase
  Urinary samples

SECONDARY OUTCOMES:
Change in sleep quality measured using the Pittsburgh Sleep Quality Index (PSQI) | Change between treatment conditions in PSQI score at treatment day 15
  A self-rated 19-item questionnaire, each of which has a range of 0 (no difficulty) to 3 (severe difficulty) points.These 19 items are combined to form 7 component scores reflecting different aspects of sleep quality. The 7 component scores are then added to yield one global score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all area.
Nocturnal skin temperature | Change between treatment conditions at bedtime at treatment days 14-15
  Skin measured around the nocturnal sleep periods

CONTACTS AND LOCATIONS:
Overall Officials: Diane B Boivin, MD, PhD, Principal Investigator — Douglas Hospital Research Centre
Locations (1):
- Centre for Study and Treatment of Circadian Rhythms, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No